CLINICAL TRIAL: NCT06311240
Title: Chronic Pain in Patients With Chronic Kidney Disease in Hemodialysis
Brief Title: Chronic Pain in Patients in Hemodialysis
Acronym: DolERC
Status: Recruiting | Type: Observational
Sponsor: Cardenal Herrera University (Other)
Collaborators: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Eva Segura Ortí, Principal Investigator, Cardenal Herrera University
Other Study IDs: 02-24-108-003
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Chronic Pain; Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Chronic Pain
MeSH Terms: conditions — Chronic Pain; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Salivary Cortisol: Physiological stress assessment will be performed simply by measuring cortisol levels in a saliva sample and subsequently analyzed using the ELISA method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participant with CKD: Participant with CKD answering the questionnaires

SUMMARY:
Pain is one of the most common symptoms among patients with End Stage Renal Disease (ESRD), and often goes unrecognized or inadequately managed in hemodialysis patients. More than 50% of patients undergoing hemodialysis suffer from pain, with 75% of them being treated ineffectively due to healthcare professionals' lack of awareness of this symptom. Therefore, pain management in this population is a complex and challenging task for healthcare providers. The most prevalent pain syndromes in hemodialysis patients include musculoskeletal disorders, metabolic neuropathies, in addition to typical intradialytic pain.

The aim of this study is to assess the presence and characteristics of chronic pain in patients with ESRD undergoing hemodialysis to determine whether it is relevant to include the management of chronic pain in the holistic treatment (physical activity, nutrition, and psychological support) already being implemented in various studies for these patients.

DETAILED DESCRIPTION:
Chronic Kidney Disease (CKD) has an estimated prevalence ranging from 13.4% to 10.6% across stages 1 to 5. These data indicate that CKD is recognized as a major global health issue, with high healthcare costs. Its incidence increases with age, with individuals over 65 years old comprising 40% of CKD patients. Gender differences exist, with males being more affected, although females exhibit greater frailty and severity. This population often presents high comorbidity with other conditions such as diabetes, hypertension, and cardiovascular diseases, along with malnutrition, sedentary lifestyles, poor health-related quality of life, low functional capacity, frailty, high levels of dependency, and, recently evidenced, pain. All of these factors are associated with increased mortality risk, exceeding 15% annually. Cardiovascular disease is the leading cause of death in patients with advanced CKD and a significant risk factor for peripheral arterial disease and lower limb amputation.

Chronic pain imposes a significant personal and economic burden, affecting over 30% of people worldwide. Unlike acute pain, which serves a protective function, chronic pain may be better considered as a disease itself, with both physical and psychological implications. There has been a growing acceptance of the biopsychosocial model in addressing patients with chronic pain, understanding pain as "an unpleasant sensory and emotional experience associated with actual or potential tissue damage, or described in terms of such damage," according to the International Association for the Study of Pain (IASP). This perspective considers pain not only as a purely nociceptive experience but also as a personal experience involving both biological and emotional/psychological components.

Pain is one of the most common symptoms among patients with end-stage CKD, often going unrecognized or inadequately managed. Barriers to proper pain management include limited awareness of the problem, inadequate medical education, and common misconceptions about the inevitability of pain in older adults and HD patients. More than 50% of hemodialysis patients suffer from pain, with 75% of them receiving ineffective treatment due to healthcare professionals' lack of awareness of this symptom. Therefore, pain management in this population is a complex and challenging task. The most prevalent pain syndromes in hemodialysis patients include musculoskeletal disorders, metabolic neuropathies, and typical intradialytic puncture pain.

Patients with chronic pain from musculoskeletal disorders have been shown to exhibit high levels of catastrophizing, fear of movement, anxiety, depression, sleep disturbances, and elevated salivary cortisol levels due to the stress caused by chronic pain and the prevalence of musculoskeletal disorders as potential causes of pain in CKD patients.

Hormonal alterations at the hypothalamic-pituitary axis (HPA) level are frequently observed with worsening renal function. Traditionally, these alterations have been understood as a consequence of renal insufficiency. However, recent evidence suggests the involvement of such hormonal disorders in the genesis of CKD. The HPA axis controls stress responses through a negative feedback mechanism. If chronic pain is considered a stressor, a reciprocal response is triggered, with increased pain activating physiological mechanisms responding to stress, such as elevated cortisol, thereby increasing perceived pain. Chronic pain induces a chronic increase in cortisol and other central mediators of the HPA axis. Cortisol is one of the physiological indices used to quantify stress, with salivary cortisol levels reflecting HPA axis activity and quantifiable non-invasively through saliva samples using ELISA methods. Currently, physiological stress assessment is easily performed by measuring cortisol levels in saliva samples.

There is a gap in the literature regarding this topic as it has not been studied whether patients with advanced-stage CKD undergoing hemodialysis present the same characteristics of chronic pain as other pathologies, such as musculoskeletal disorders.

Methodology Study Type: A cross-sectional observational study will be conducted. Since no previous studies exist, a study with n: 20 will be conducted, and based on this data, the sample size calculation will be performed. Randomization and blinding will not be performed, and no intervention is planned.

Variables

The following measurement variables will be used in this study:

Biomarkers:

* Salivary Cortisol: Physiological stress assessment will be performed simply by measuring cortisol levels in a saliva sample and subsequently analyzed using the ELISA method.

The following questionnaires will be used to measure health condition variables:

* Sleep Quality: The validated Spanish version of the Pittsburgh Sleep Quality Index will be used.
* Stress: The validated Spanish version of the Perceived Stress Questionnaire will be used.
* Disease Self-Management: The self-efficacy questionnaire will be used.

The following questionnaire and physical variable measurement will be used to measure variables related to chronic pain:

* Chronic Pain Severity Scale: The validated Spanish version of the Chronic Pain Severity Scale will be used.
* Pressure Pain Thresholds (PPT): This variable is used to assess if the patient presents symptoms compatible with central sensitization. Pressure will be applied with an algometer at two bilateral points, the second rib and knee. Each measured subject will be instructed to say 'stop' when the pressure sensation becomes the first sensation of pain. Each measurement will be repeated three times with 10 seconds of rest between them.

The following questionnaire will be used to measure headache-related variables:

* HIT-6: The validated Spanish version of the Headache Impact Test-6 questionnaire will be used.

The following questionnaires will be used to measure behavioral variables:

* Catastrophizing: The validated Spanish version of the Pain Catastrophizing Scale will be used.
* Anxiety and Depression: The validated Spanish version of the Hospital Anxiety and Depression Scale (HADS) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients with End-Stage Renal Disease (ESRD)
* Have been on hemodialysis treatment for at least 3 months and are medically stable.
* Able to walk a few steps, even if they require walking aids such as canes or walkers.

Exclusion Criteria:

* Myocardial infarction in the past 6 weeks.
* Unstable angina during exercise or at rest.
* Amputation of lower limbs above the knee without prosthetics.
* Cerebrovascular disease such as stroke or transient ischemic attacks in the last 6 months or with significant sequelae affecting lower limb mobility.
* Musculoskeletal or respiratory disorders that worsen with exercise.
* Inability to perform study tests/questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients selected by Nephrologists in different Hemodialysis units collaborating in the current project, which includes holistic treatment through non-immersive virtual reality both at the dialysis center and at home, will be invited to participate in this study. Patients from different Hemodialysis units (Hospital de Manises and with approval from the Clinical Research Ethics Committee (CEIC) at the Consorcio Sanitario de Terrassa) and patients who are part of the renal patient association ALCER España (Association for the Fight against Kidney Diseases) will also be selected.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Stress level assessed by the salivary cortisol test | Baseline
  Higher stress present higher cortisol levels
Stress level assessed by the perceived stress scale (PSS) | Baseline
  The minimal score is 0. The maximum PSS score is 56. The higher score obtained, the higher stress level

SECONDARY OUTCOMES:
Self- efficacy assessed by questionnaire | Baseline
  The minimal score is 0. The maximun Self-efficacy score is 40. The lower score obtained , the lower self-efficacy
Quality of sleep assessed by Pittsburgh Sleep Quality Index | Baseline
  The minimal score is 0. The maximun quality index score is 21. The higher score obtained, the lower quality of sleep
The impact of headaches on life assessed by Headache Impact Test-6 | Baseline
  The minimal score is 0. The maximun Headache Impact Test-6 score is 79. The higher score obtained, the higher impact of headaches on life
Anxiety and depression assessed by Hospital anxiety and depression scale (HADS) | Baseline
  The minimal score is 0. The cutoff point for the two subscales, anxiety and depression, is 8 and < 10. The higher score obtained, The higher impact of anxiety and depression levels on life.
Aspects of catastrophic cognitions about pain-rumination, magnification, and helplessness assessed by The Pain Catastrophizing Scale (PCS) | Baseline
  The minimal score is 0. The maximun The Pain Catastrophizing Scale score is 52. The higher score obtained, the higher impact of pain rumination, magnification and helplessness on life related to pain.
Chronic pain assessed by Chronic Pain Grade Questionnaire | Baseline
  The minimal score is 0. The maximun Chronic Pain Grade Questionnaire score is 70. The higher score obtained, the higher impact of chronic pain on life

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Garrigós-Pedrón, PhD, Principal Investigator — Universidad Cardenal Herrera-CEU, CEU Universities
Locations (2):
- Spain (2):
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Universidad Cardenal Herrera-CEU, CEU Universities, Alfara del Patriarca, Valencia

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared under request

REFERENCES:
- [Background] Hill NR, Fatoba ST, Oke JL, Hirst JA, O'Callaghan CA, Lasserson DS, Hobbs FD. Global Prevalence of Chronic Kidney Disease - A Systematic Review and Meta-Analysis. PLoS One. 2016 Jul 6;11(7):e0158765. doi: 10.1371/journal.pone.0158765. eCollection 2016. PMID 27383068
- [Background] Costa YM, Porporatti AL, Stuginski-Barbosa J, Bonjardim LR, Speciali JG, Conti PC. Headache attributed to masticatory myofascial pain: impact on facial pain and pressure pain threshold. J Oral Rehabil. 2016 Mar;43(3):161-8. doi: 10.1111/joor.12357. Epub 2015 Oct 6. PMID 26440358
- [Background] Cohen SP, Vase L, Hooten WM. Chronic pain: an update on burden, best practices, and new advances. Lancet. 2021 May 29;397(10289):2082-2097. doi: 10.1016/S0140-6736(21)00393-7. PMID 34062143
- [Background] Hylands-White N, Duarte RV, Raphael JH. An overview of treatment approaches for chronic pain management. Rheumatol Int. 2017 Jan;37(1):29-42. doi: 10.1007/s00296-016-3481-8. Epub 2016 Apr 23. PMID 27107994
- [Background] Coluzzi F. Assessing and Treating Chronic Pain in Patients with End-Stage Renal Disease. Drugs. 2018 Sep;78(14):1459-1479. doi: 10.1007/s40265-018-0980-9. PMID 30206801
- [Background] Raina R, Krishnappa V, Gupta M. Management of pain in end-stage renal disease patients: Short review. Hemodial Int. 2018 Jul;22(3):290-296. doi: 10.1111/hdi.12622. Epub 2017 Dec 11. PMID 29227577
- [Background] Luque-Suarez A, Martinez-Calderon J, Falla D. Role of kinesiophobia on pain, disability and quality of life in people suffering from chronic musculoskeletal pain: a systematic review. Br J Sports Med. 2019 May;53(9):554-559. doi: 10.1136/bjsports-2017-098673. Epub 2018 Apr 17. PMID 29666064
- [Background] Sole E, Racine M, Tome-Pires C, Galan S, Jensen MP, Miro J. Social Factors, Disability, and Depressive Symptoms in Adults With Chronic Pain. Clin J Pain. 2020 May;36(5):371-378. doi: 10.1097/AJP.0000000000000815. PMID 32040011
- [Background] Fujiwara A, Ida M, Watanabe K, Kawanishi H, Kimoto K, Yoshimura K, Shinohara K, Kawaguchi M. Prevalence and associated factors of disability in patients with chronic pain: An observational study. Medicine (Baltimore). 2021 Oct 8;100(40):e27482. doi: 10.1097/MD.0000000000027482. PMID 34622878
- [Background] Meuwese CL, Carrero JJ. Chronic kidney disease and hypothalamic-pituitary axis dysfunction: the chicken or the egg? Arch Med Res. 2013 Nov;44(8):591-600. doi: 10.1016/j.arcmed.2013.10.009. Epub 2013 Nov 8. PMID 24215784
- [Background] Arregger AL, Cardoso EM, Tumilasci O, Contreras LN. Diagnostic value of salivary cortisol in end stage renal disease. Steroids. 2008 Jan;73(1):77-82. doi: 10.1016/j.steroids.2007.09.001. Epub 2007 Sep 11. PMID 17945323
- [Background] Reyes del Paso GA, Perales Montilla CM. Haemodialysis course is associated to changes in pain threshold and in the relations between arterial pressure and pain. Nefrologia. 2011;31(6):738-42. doi: 10.3265/Nefrologia.pre2011.Oct.10902. English, Spanish. PMID 22130291